CLINICAL TRIAL: NCT07327684
Title: Research on the Morphology and Functional Assessment of Brown Adipose Tissue With Photoacoustic Imaging
Brief Title: Photoacoustic/Ultrasound Imaging of Brown Adipose Tissue Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PA/US Brown Adipose Tissue
Record Dates: First submitted 2025-11-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Insulin Resistance; Metabolic Syndrome
Keywords: Metabolic syndrome; Insulin resistance; Brown adipose tissue; Photoacousitc imaging
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brown adipose tissue assessment of healthy volunteers based on PA/US imaging (Experimental): Establish a non-invasive, real-time PAI method for quantitative characterization of human BAT morphology and metabolic function and evaluate the baseline of BAT PA parameters in healthy population.
  Interventions: Device: Multi-wavelength PA/US imaging scanning and cold exposure
- Brown adipose tissue assessment of patients with metabolic syndrome based on PA/US imaging (Experimental): Evaluate the BAT PA parameters in patients with metabolic syndrome.
  Interventions: Device: Multi-wavelength PA/US imaging scanning and cold exposure

INTERVENTIONS:
Device: Multi-wavelength PA/US imaging scanning and cold exposure — Participants will undergo multi-wavelength PAI scans of BAT region under normal conditions and after 30-60 mins cold exposure to assess BAT activation.
  Arms: Brown adipose tissue assessment of healthy volunteers based on PA/US imaging
Device: Multi-wavelength PA/US imaging scanning and cold exposure — Participants will undergo multi-wavelength PAI scans of BAT region under normal conditions and after 30-60 mins cold exposure to assess BAT activation.
  Arms: Brown adipose tissue assessment of patients with metabolic syndrome based on PA/US imaging

SUMMARY:
The goal of this study is to develop a novel, non-invasive, real-time photoacoustic imaging (PAI) technology for quantifying brown adipose tissue (BAT) and to investigate the differences in BAT morphology and metabolic function between healthy individuals and patients with metabolic syndrome.

The main questions it aims to answer are:

1. Can PAI technology quantify BAT metabolic function and establish standardized PAI parameters for BAT assessment?
2. Can PAI parameters distinguish the BAT characteristics of healthy volunteers from patients with metabolic syndrome?

Both healthy adults and patients diagnosed with metabolic syndrome will be recruited. Participants will undergo PAI scans of BAT region under normal conditions and after cold exposure to assess BAT activation.

The ultimate goal is to validate this radiation-free PAI method as a convenient and effective tool for evaluating BAT metabolism, potentially aiding in early diagnosis and treatment monitoring of metabolic syndrome.

DETAILED DESCRIPTION:
Brown adipose tissue (BAT) is a thermogenic organ that plays a beneficial role in whole-body metabolism by burning calories to generate heat. Its activity is inversely associated with obesity, insulin resistance, and metabolic syndrome. A key challenge in advancing BAT research and its clinical translation is the lack of a non-radiative, non-invasive imaging technique suitable for repeated use in both healthy and diseased populations. The current gold standard, [¹⁸F]FDG-PET/CT, involves ionizing radiation, limiting its application in longitudinal studies and healthy volunteer screening.

Photoacoustic imaging (PAI) is an emerging hybrid modality that combines high optical contrast with deep ultrasound penetration. It can uniquely quantify tissue composition by detecting intrinsic contrasts like lipids and hemoglobin, making it ideally suited for assessing BAT's lipid content, blood perfusion and vascular oxygenation, which are key aspects of its metabolic function.

The objectives of this study are:

1. To develop and technically optimize a non-invasive, real-time PAI protocol for quantitative characterization of human BAT morphology and metabolic function.
2. To establish a set of standardized, quantitative PAI parameters (e.g., related to blood perfusion, lipid composition, blood oxygen saturation) for BAT assessment.
3. To compare the baseline PAI parameters of BAT between healthy volunteers and patients with metabolic syndrome.

Both healthy control group and the patient group will be recruited to undergo PAI scans targeting the supraclavicular BAT depots. All scans will be performed under normal conditions and a standardized cold exposure protocol to stimulate BAT activity. Quantitative PAI parameters (e.g., total hemoglobin, lipid concentration, oxygen saturation) will be extracted and compared between the Healthy Control group and the Patient group using appropriate statistical tests.

This study will not only develop a novel PAI technology for BAT imaging but also utilize it to directly investigate a critical biological question: how BAT differs between health and disease. By establishing PAI-based biomarkers that can distinguish these states, this research aims to provide a powerful, radiation-free tool for the early detection of metabolic dysfunction, risk stratification, and objective monitoring of therapeutic efficacy for insulin resistance and related metabolic syndrome.

ELIGIBILITY:
Criteria for Healthy Subjects:

(INCLUSION CRITERIA)

1. Healthy individuals over 18 years of age.
2. Body Mass Index (BMI) < 30.
3. No history of metabolic diseases, rheumatic immune diseases, or cardiovascular and cerebrovascular diseases.
4. Not currently using any sympathomimetic or sympatholytic drugs.
5. Non-smoker and does not consume excessive alcohol.

(EXCLUSION CRITERIA)

1. Weight change > 5% within 3 months prior to enrollment.
2. BMI ≥ 30.
3. Diagnosis of metabolic disease, rheumatic immune disease, cardiovascular and cerebrovascular disease, or malignant tumor.
4. Use of sympathomimetic or sympatholytic drugs within 3 months prior to enrollment.
5. Smoker or consumes excessive alcohol.
6. Diagnosis of Raynaud's disease, or intolerance/allergy to cold stimulation.
7. Currently pregnant, lactating, or menstruating.
8. Contraindications to the injection of the radionuclide tracer Fluorodeoxyglucose (18F-FDG) or other conditions unsuitable for PET-CT examination.

Criteria for Patients with Metabolic Syndrome and Insulin Resistance-Related Diseases:

(INCLUSION CRITERIA)

1. Age between 18 and 60 years.
2. Must meet 3 or more of the following criteria:

   1. Waist circumference ≥ 90 cm for males, ≥ 85 cm for females.
   2. Fasting blood glucose ≥ 6.10 mmol/L (110 mg/dl) OR 2-hour postprandial blood glucose ≥ 7.80 mmol/L (140 mg/dl) OR previously diagnosed diabetes.
   3. Blood pressure ≥ 130/85 mmHg OR previously diagnosed hypertension and under treatment.
   4. Fasting triglycerides (TG) ≥ 1.7 mmol/L (150 mg/dl).
   5. Fasting high-density lipoprotein cholesterol (HDL-C) < 1.0 mmol/L (40 mg/dl).
3. Patients diagnosed with Polycystic Ovary Syndrome (PCOS), defined as meeting two or more of the following criteria and excluding other endocrine diseases that could cause similar symptoms: hyperandrogenism, ovulatory dysfunction, polycystic ovary morphology.

(EXCLUSION CRITERIA)

1. Diagnosis of Type 1 diabetes or other specific types of diabetes.
2. Presence of acute diabetic complications or severe chronic diabetic complications.
3. History of acute or chronic pancreatitis, or pancreatic tumors.
4. Heart failure, unstable angina, myocardial infarction within the past 12 months, cerebral infarction, severe arrhythmia, or severe hypertension (blood pressure > 180/110 mmHg despite antihypertensive medication).
5. Severe hepatic or renal dysfunction.
6. Comorbid malignant tumors or other severe chronic diseases.
7. Received glucose-lowering therapy within 3 months prior to enrollment OR a total of more than 3 months of glucose-lowering therapy in the past 2 years.
8. Diagnosis of rheumatic immune diseases.
9. Diagnosis of Raynaud's disease, or intolerance/allergy to cold stimulation.
10. Currently pregnant, lactating, or menstruating.
11. Contraindications to the injection of the radionuclide tracer Fluorodeoxyglucose (18F-FDG) or other conditions unsuitable for PET-CT examination.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in photoacoustic imaging (PAI)-derived total hemoglobin concentration within brown adipose tissue (BAT) after cold exposure. | Baseline and immediately after a standardized 0.5-1 hour cold exposure procedure
  The concentration of total hemoglobin (a.u.) within the BAT region of interest will be measured using a co-registered photoacoustic and ultrasound (PA/US) imaging system. The change (Δ) will be calculated as the value after a standardized cold exposure divide the value at baseline.
Change in photoacoustic imaging (PAI)-derived lipid concentration within brown adipose tissue (BAT) after cold exposure | Baseline and immediately after a standardized 0.5-1hour cold exposure procedure.
  The lipid concentration (a.u.) within the BAT region of interest will be measured using a co-registered photoacoustic and ultrasound (PA/US) imaging system. The change (Δ) will be calculated as the value after a standardized cold exposure minus the value at baseline.
Change in photoacoustic imaging (PAI)-derived oxygen saturation within brown adipose tissue (BAT) after cold exposure | Baseline and immediately after a standardized 0.5-1 hour cold exposure procedure.
  The oxygen saturation (in %) within the BAT region of interest will be measured using a co-registered photoacoustic and ultrasound (PA/US) imaging system. The change (Δ) will be calculated as the value after a standardized cold exposure minus the value at baseline.
Difference between healthy volunteers and patients with metabolic syndrome in the cold-induced change of photoacoustic imaging (PAI)-derived total hemoglobin concentration within brown adipose tissue (BAT). | Through study completion, an average of 24 months.
  The change (Δ) in total hemoglobin concentration (a.u.) after cold exposure (as defined in Outcome 1) will be compared between healthy volunteers and patients diagnosed with metabolic syndrome.
Difference between healthy volunteers and patients with metabolic syndrome in the cold-induced change of photoacoustic imaging (PAI)-derived lipid concentration within brown adipose tissue (BAT) | Through study completion, an average of 24 months
  The change (Δ) in lipid concentration (a.u.) after cold exposure (as defined in Outcome 2) will be compared between healthy volunteers and patients diagnosed with metabolic syndrome.
Difference between healthy volunteers and patients with metabolic syndrome in the cold-induced change of photoacoustic imaging (PAI)-derived oxygen saturation within brown adipose tissue (BAT) | Through study completion, an average of 24 months
  The change (Δ) in oxygen saturation (in %) after cold exposure (as defined in Outcome 3) will be compared between healthy volunteers and patients diagnosed with metabolic syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China